CLINICAL TRIAL: NCT02235467
Title: Multisite Study: Acquisition of Social Skills in Children With Autism Using Video Modeling in Parental Training
Brief Title: Multisite Study: Parental Training Using Video Modelling to Develop Social Skills in Children With Autism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Mackenzie Presbiterian University, São Paulo, Brazil (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jair Mari, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1157-8984; 2012/51584-0 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Autism Spectrum Disorders
Keywords: autism; videomodeling; behavioral therapy; parental training
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABA parent training (Active Comparator): Applied Behavior Analysis parent training using videomodeling in 21 sessions
  Interventions: Behavioral: ABA parent training
- ABA parent training control (No Intervention)

INTERVENTIONS:
Behavioral: ABA parent training — A parent training based on Applied Behavior Analysis that is going to be delivered by video modeling in 21 weeks
  Other Names: Applied Behavior Analysis parent training using videomodeling
  Arms: ABA parent training

SUMMARY:
This is a Brazilian multisite study to test the efficacy of an Applied Behavior Analysis (ABA) parent training using video modeling to teach parents of children with Autism techniques to apply to their children in order to improve eye contact and joint attention behaviors.

Our hypothesis is that children with Autism whose parents will be trained by videomodeling will have better eye contact and joint attention behaviors compared to children with Autism whose parents will not be trained.

DETAILED DESCRIPTION:
Applied Behavior Analysis (ABA) is an intervention with proven efficacy in treating impairments on social functioning and daily-life activities of individuals with Autism Spectrum Disorder (ASD). In Brazil we have a limited number of qualified professionals and an increasing demand of families non-served in the public health system.

Our main objective is to standardize and test the efficacy of a model for parent training using video modeling for teaching eye contact and joint attention behaviors in children with ASD. These two behaviors are essential to develop adequate social interaction, the core impaired domain in ASD. It is a multisite study to be carried out at the Universidade Federal de São Paulo, Universidade de São Paulo and Universidade Presbiteriana Mackenzie. The sample will be composed of 70 children divided in control and intervention groups that will be randomly chosen. The intervention should be carried out in 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Autism Spectrum Disorders
* Diagnosis of Autism Spectrum Disorders by means of ADI
* IQ equal or lower than 70 by means of SON
* Main caregiver's level of education > primary education

Exclusion Criteria:

* IQ lower than 50 by means of SON
* Child who is receiving ABA therapy at least 10 hours per week
* Main caregiver diagnosed with Autism Spectrum Disorders

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Acquisition from baseline of new behaviors at 8 weeks | baseline assessment to 8 weeks of therapy
  acquisition of new behaviors (eye contact and joint attention) checked through taped interactions between child and a family member
Acquisition from baseline of new behaviors at 16 weeks | baseline assessment to 16 weeks
  acquisition of new behaviors (eye contact and joint attention) checked through taped interactions between child and a family member
Acquisition from baseline of new behaviors at 21 weeks | baseline to 21 weeks
  acquisition of new behaviors (eye contact and joint attention) checked through taped interactions between child and a family member

SECONDARY OUTCOMES:
Change from baseline in Eye-tracking at 21 weeks | baseline assessment to 21 weeks
  Latency, duration, and sequence of visual fixations measured with eye-tracking
Change from baseline in Vineland Scale at 21 weeks | baseline assessment to 21 weeks
  Adaptative behavior using Vineland Scale
Change from baseline in SON-R 2½-7 at 21 weeks | baseline assessment to 21 weeks
  Improve on SON-R 2½-7 that is an intelligence coefficient test developed for deaf people
Change from baseline in Zaritt Burden Interview at 21 weeks | baseline assessment to 21 weeks
  The Zaritt Burden Interview measures the caregiver burden of taking care of the relative with psychiatric disorder
Change from baseline in OERA at 21 weeks | baseline assessment to 21 weeks
  OERA (Observação Estruturada para Rastreamento de Autismo) is a taped structured observation to screen Autism that was developed by Brazilian researchers.

OTHER OUTCOMES:
Change from baseline in KAP at 21 weeks | baseline assessment to 21 weeks
  Improvement on the knowledge, attitude and practice (KAP) questionnaire
Change from baseline in Hamilton scalels and at 21 weeks | baseline assessment to 21 weeks
  Improvement on the Hamilton Depression and Anxiety scales of the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Sheila C Caetano, MD, PhD, Study Director — Federal University of São Paulo, São Paulo, Brazil
Locations (1):
- Federal University of São Paulo Department of Psychiatry, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Correia BSB, de Moraes Pontes JG, Nani JVS, Villalta F, Mor NC, Bordini D, Brunoni D, Brentani H, Mari JJ, Hayashi MAF, Tasic L. 1H NMR Metabolomics and Lipidomics To Monitor Positive Responses in Children with Autism Spectrum Disorder Following a Guided Parental Intervention: A Pilot Study. ACS Chem Neurosci. 2023 Mar 15;14(6):1137-1145. doi: 10.1021/acschemneuro.2c00735. Epub 2023 Feb 21. PMID 36808953